CLINICAL TRIAL: NCT04309513
Title: Evaluation of the Personal Activity Intelligence (PAI) Score in a Corporate Wellness Setting.
Brief Title: Evaluation of the Personal Activity Intelligence (PAI) Score
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: Memorial Health System (Other)
Responsible Party: Principal Investigator, David Drozek, Associate Professor, Ohio University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20-X-88
Record Dates: First submitted 2020-03-11; First posted 2020-03-16 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step Counter to motivate physical activity (Active Comparator): Participants will be encouraged to work up to achieving at least 10,000 steps a day, higher if possible and reasonable, as measured by a wearable device.
  Interventions: Behavioral: Step Counter to motivate physical activity
- PAI score to motivate physical activity (Experimental): Participants will be encouraged to work up to and maintain the highest PAI score possible, with 100 being the ideal, as measured by a wearable device.
  Interventions: Behavioral: PAI score to motivate physical activity

INTERVENTIONS:
Behavioral: PAI score to motivate physical activity — Participants will be encouraged to work up to and maintain the highest PAI score possible, with 100 being the ideal, as measured by a wearable device. Their devices and an accompanying app will provide them with an ongoing real time calculation of the PAI score.
  Arms: PAI score to motivate physical activity
Behavioral: Step Counter to motivate physical activity — Step Counter to motivate physical activity
  Arms: Step Counter to motivate physical activity

SUMMARY:
This will be a prospective randomized controlled study to evaluate the effectiveness of the Personal Activity Intelligence (PAI) Score to encourage physical activity.

Participants will utilize a wearable wrist device that will provide data pertaining to physical activity, to include steps taken, miles walked, heart rate, calories burned, etc. The intervention group devices will also provide a visible PAI score and will be given information about a PAI app they can install on their smart phone to monitor their activity

Control participants will be encouraged to work up to at least 10,000 steps a day, higher if possible and reasonable.

Those with a device that displays a PAI score (study participants) will be encouraged to work up to and maintain the highest PAI score possible, with 100 being the ideal.

DETAILED DESCRIPTION:
The objective is to determine if utilizing the PAI score as a single measure for goal setting is superior to monitoring steps / distance, calories burned, and / or time in aerobic activity in achieving improvements in health.

Study participants will have enrolled in Corporate Wellness Program at Memorial health System (MHS), and have met the inclusion criteria and consented.

Participants will be randomly assigned to one of the groups. Members from the same household will be assigned to the same group together.

All devices will be linked, via smart phone, to a fitness tracker app that is imbedded in the MHS medical record, and has a patient access portal accessible to the patient via website or app on a smart phone or tablet.

The intervention device will also link to a smart phone app developed by PAI that displays PAI score to the participant as well as other data, to allow tracking.

Participants will be asked to wear their devices on at least two nights during the first week, and daily while awake, except when bathing for the next 12 weeks.

Participants, having enrolled in the wellness program, will already, as a part of that study, have agreed to have data collected at baseline and yearly thereafter, including BMI, blood pressure, resting pulse, lipid panel, hemoglobin A1c, health risk assessment survey, absenteeism and health claims data at baseline and yearly thereafter. If not collected within 60 days, a new set of data will be collected to serve as baseline for this study. Specifically for this study this data collection (including lab analysis) will also be repeated at 12 weeks and 6 months. All blood draws will be done at any MHS lab, by qualified phlebotomists, according to standard hospital policy.

The control group will be asked to work toward a goal of at least 10,000 steps a day, which can be seen on their device, as well as on the accompanying app.

The intervention group will be encouraged to work up to and maintain the highest PAI score possible, with at least 100 being the ideal. PAI will provide weekly summary data on participants that will allow additional evaluation correlating level of physical activity / PAI score with participant results. This data will be reported with a participant code. PAI will provide a master code linking the participant code to an email address for correlation of all data for analysis. This master code will be maintained on an encrypted device.

ELIGIBILITY:
Inclusion Criteria:

* Adult who is enrolled in the Memorial Health System (MHS) corporate wellness study.
* Is interested in increasing level of physical activity.
* Is able to walk at least a mile a day.
* Has a device that is compatible with the software (Apple watch, Fitbit, Garmin) or is willing to purchase a device for $25 offered as part of this study.

Exclusion Criteria:

* Does not speak English
* Has been told by a medical provider to not participate in physical activity.
* Is taking a beta blocker medication (which slows the heart rate) (https://www.medicinenet.com/beta_blockers/article.htm#list_of_examples_of_brand_and_generic_names_for_beta_blockers_available)
* Has a medical condition that prevents walking at least a mile a day.
* Has a pacemaker or defibrillator.
* Is currently in cardiac rehab
* Is not able to manage an app on a "smart phone".
* Deemed unsuitable to the program by Dr. Drozek or other members of the wellness team. (mental impairment, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Physical Activity Level | 2 years
  Change in Exercise Vital Signs obtained by survey at 2 years.
  1. Are you able to walk a mile without significant pain or discomfort? ❒ Yes ❒ No
  2. In the past 7 days, how many days did you exercise? ______ days
  3. On days when you exercised, for how long did you exercise (in minutes)?
     ❒______ minutes per day
     ❒ Does not apply
  4. How intense was your typical exercise?
     * Light (like stretching or slow walking)
     * Moderate (like brisk walking)
     * Heavy (like jogging or swimming)
     * Very heavy (like fast running or stair climbing)
     * I am currently not exercising

SECONDARY OUTCOMES:
Daily Step Count | 2 years
  Change in number of steps per day achieved at 2 years
BMI | 2 years
  Change in body mass index at 2 years, calculated by measuring height in feet / inches and weight in pounds.
Glycosylated Hemoglobin (HbA1c) | 2 years
  Change in % of HbA1c from baseline at 2 years.
Total cholesterol | 2 years
  Change in mg/dl from baseline at 2 years.
Low Density Lipoprotein (LDL) cholesterol | 2 years
  Change in mg/dl from baseline at 2 years.
High Density Lipoprotein (HDL) cholesterol | 2 years
  Change in mg/dl from baseline at 2 years.
Triglycerides | 2 years
  Change in mg/dl from baseline at 2 years.
Blood pressure (systolic and diastolic) | 2 years
  Change in blood pressure in mm Hg from baseline at 2 years.
Mood | 2 years
  Change From baseline in mood scores on the The Patient Health Questionnaire-4 (PHQ-4) at 2 years, Higher score is more abnormal

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided